CLINICAL TRIAL: NCT00616148
Title: Pharmacodynamic Evaluation of YKP3089 in Epilepsy Patients With a Photo-induced Paroxysmal EEG-Response: Proof of Principle
Brief Title: Efficacy of YKP3089 in Patients With Photosensitive Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Collaborators: The Epilepsy Study Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA40616
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Cenobamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- YKP3089 (Experimental)
  Interventions: Drug: YKP3089

INTERVENTIONS:
Drug: YKP3089 — Oral dosage form
  Arms: YKP3089
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the ability of a single oral dose of YKP3089 to abolish or clearly reduce the IPS-induced photo-paroxysmal EEG response in photosensitive epilepsy patients, and to measure the onset and duration of the effect. Several cohorts will be used, to sequentially investigate different doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-60 years.
* A diagnosis and history of epilepsy for which patients are on 0-2 concomitant antiepileptic drugs.
* If the patient is taking two concomitant medications, the second drug must be levetiracetam, gabapentin or pregabalin.
* A reproducible IPS-induced photo-paroxysmal response (PPR) on EEG of at least 3 points on a frequency assessment scale (See Section 6.16) in at least one eye condition and no change of more than 3 frequencies in 2 repeated measurements recorded over the 2 months prior to study entry in at least one eye condition.
* Patients in otherwise good health (with the exception of epilepsy), as determined by the PI via the medical history, a physical examination and screening laboratory investigations.
* A body mass index (BMI) between 18 and 35.
* Able and willing to provide written informed consent to participate in the study in accordance with the ICH, GCP guidelines.

Exclusion Criteria:

* A history of non epileptic seizures (e.g. metabolic, structural or pseudo-seizures).
* Women who are pregnant or lactating.
* Women of reproductive potential who do not agree to use effective birth-control methods.
* Patients taking medications that are known substrates of CYP2B6 and CYP2C19 including but not limited to phenytoin, Phenobarbital, omeprazole, fluvoxamine and efavirenz.
* Any clinically significant laboratory abnormality which, in the opinion of the investigator, will exclude the patient from the study.
* An active CNS infection, demyelinating disease, degenerative neurological disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
* Any clinically significant psychiatric illness, psychological or behavioral problems which, in the opinion of the investigator, would interfere with the patient's ability to participate in the study.
* Patients who are suffering from clinically significant active liver disease, porphyria or with a family history of severe hepatic dysfunction indicated by abnormal liver function tests greater than 3 times the upper limit of normal (AST and ALT).
* A history of alcoholism, drug abuse, or drug addiction (within the past 12 months).
* Patients who would normally be contraindicated for YKP3089 administration.
* Patients who have participated in any other trials involving an investigational product or device within 30 days of screening or longer as required by local regulations.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Determine if YKP3089 will reduce or abolish the photosensitivity response as compared to placebo. | At the completion of each cohort

SECONDARY OUTCOMES:
Assessment of serum concentrations of concomitant AEDs during administration of YKP3089 as compared to the placebo day. Assessment of safety/tolerability at multiple dose levels. | At the completion of each cohort

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline French, M.D., Principal Investigator — NYU MEDICAL CENTER
Locations (4):
- United States (4):
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Cornell Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Pennsylvania Epilepsy Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Kasteleijn-Nolst Trenite DGA, DiVentura BD, Pollard JR, Krauss GL, Mizne S, French JA. Suppression of the photoparoxysmal response in photosensitive epilepsy with cenobamate (YKP3089). Neurology. 2019 Aug 6;93(6):e559-e567. doi: 10.1212/WNL.0000000000007894. Epub 2019 Jul 10. PMID 31292226